CLINICAL TRIAL: NCT02506517
Title: Molecular Basket Trial In Multiple Malignancies With Common Target Pathway Aberrancies
Brief Title: A Study of Afatinib in Patients With Advanced Cancer With Changes in the HER Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOBILITY-003
Record Dates: First submitted 2015-07-15; First posted 2015-07-23 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumors
Keywords: HER pathway aberrations
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (Experimental): Afatinib, orally, at a dose of 40 mg once a day, every day of each 28 day cycle.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib
  Other Names: GIOTRIF

SUMMARY:
This is a phase 2 study (the second phase in testing a new drug) to see how useful an investigational drug called afatinib is in patients with advanced cancer with changes in the HER gene.

Afatinib is a drug that is approved by Health Canada for the treatment of advanced lung cancer with changes in the HER gene. Afatinib works by attaching to and blocking a protein called HER from working. HER is an important protein that contributes to the growth of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have had any number of treatment lines in the curative or metastatic setting for their solid tumors.
* Age 18 years or older.
* At least one measurable lesion
* In patients with previous treatment, evidence of progression of cancer, as per the opinion of the investigator must be present
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function
* Willingness to undergo fresh tumor biopsy at certain timepoints
* Recovered from any previous therapy related side effects
* Able to provide written consent

Exclusion Criteria:

* Chemotherapy, biological therapy or investigational agents within 3 weeks prior to the start of study treatment.
* Hormonal treatment within 3 weeks prior to start of study treatment.
* Radiotherapy within 3 weeks prior to randomization with exceptions
* Major surgery within 3 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Known exposure to any epidermal growth factor receptor (EGFR), human epidermal growth factor receptor (HER) 2, HER3 or pan-HER inhibitors, such as, but not limited to afatinib or dacomitinib.
* Patients with inability to swallow whole tablets for afatinib are allowed on the study, but diluted tablets must be taken orally.
* Presence of malabsorption problems including, but not exclusively limited to chronic diarrhea and uncontrolled inflammatory bowel disease.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to study entry
* Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 28 days after treatment has ended.
* Female patients of childbearing potential who are nursing or are pregnant or are not using an acceptable method of birth control, or do not plan to continue using this method throughout the study and/or do not agree to submit to pregnancy testing required by the study.
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the study drug
* Previous or concomitant malignancies at other sites, with exceptions
* Requiring treatment with any of the prohibited concomitant medications
* Known pre-existing interstitial lung disease
* Any history or presence of poorly controlled gastrointestinal disorders.
* Known active hepatitis B, active hepatitis C infection and/or known HIV carrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete response | 2 years
Number of patients with partial response | 2 years

SECONDARY OUTCOMES:
Number of Grade 1 side effects | 2 years
Number of Grade 2 side effects | 2 years
Number of Grade 3 side effects | 2 years
Number of Grade 4 side effects | 2 years
Timeframe of Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Salawu A, Hansen AR, Spreafico A, Al-Ezzi E, Webster S, Bedard PL, Doi J, Wang L, Siu LL, Abdul Razak AR. A Phase 2 Trial of Afatinib in Patients with Solid Tumors that Harbor Genomic Aberrations in the HER family: The MOBILITY3 Basket Study. Target Oncol. 2022 May;17(3):271-281. doi: 10.1007/s11523-022-00884-z. Epub 2022 May 30. PMID 35635640